CLINICAL TRIAL: NCT01776879
Title: Speech Intelligibility of Patients With Parkinsons Disease at Different Stages of the Disease Compared to First Degree Relatives of Parkinson's Disease Patients
Brief Title: Speech Intelligibility of Patients With P D Compared to First Degree Relatives of P D Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Responsible Party: Principal Investigator, Michal Roll PhD,MBA, director rnd devision, Tel-Aviv Sourasky Medical Center
Other Study IDs: TASMC-12-TG-0556-CTIL; 0556-12 (Other: TEL AVIV MEDICAL CENTER)
Record Dates: First submitted 2012-11-13; First posted 2013-01-28 (Estimated); Last update posted 2013-01-28 (Estimated); Status verified 2013-01

CONDITIONS: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- early & advanced PD 1st degree relatives: no intervention is performed in the study
- recording speech and voice: no intervention(s) will be administered
- speech intelligibility: no intervention(s) will be administered

SUMMARY:
This study will examine speech intelligibility of early parkinson's disease (PD) patients, early PD patients and first degree relatives. The investigators hypothesis that advanced PD patients will present decreased speech intelligibility more than early PD patients. Speech intelligibility of first degree relatives will be normal.

DETAILED DESCRIPTION:
in order to achieve the study's goals objective and subjective research tools will be used.

Objective tools include measuring phonation time, diadokokinetic movements of the oral structures and acoustic analysis .

Subjective tools include self reported questionnaires.

ELIGIBILITY:
Inclusion Criteria:A

* Advanced PD patients
* Early PD patients
* First degree relatives

Exclusion Criteria:

* Patients with decreased cognitive abilities
* Patients who participate in speech therapy

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Advanced PD patients Early PD patients First degree relatives
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2013-02; Primary Completion 2013-11 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Maximum phonation time | DAY 1
  maximum phonation time will be measured after taking few measurements of sentence reading.It is an observational study that aim to collect data during DAY 1 only! day 1 for outcome measure time frames There are not pre/post measurements

SECONDARY OUTCOMES:
Diadokokinetik (DDK): production time of 10x PATAKA, 7x /P/ and 7x /t/ | DAY 1
  production time of 10x PATAKA, 7x /P/ and 7x /t/ will be measured during the examination.
  It is an observational study that aim to collect data during DAY 1 only! DAY 1 for outcome measure time frames There are not pre/post measurements

CONTACTS AND LOCATIONS:
Overall Officials: Tanya Gurevich, MD, Principal Investigator — Tel-Aviv Sourasky Medical Center

REFERENCES:
- [Background] Amir O, Ashkenazi O, Leibovitzh T, Michael O, Tavor Y, Wolf M. Applying the Voice Handicap Index (VHI) to dysphonic and nondysphonic Hebrew speakers. J Voice. 2006 Jun;20(2):318-24. doi: 10.1016/j.jvoice.2005.08.006. Epub 2005 Dec 1. PMID 16324824